CLINICAL TRIAL: NCT05462340
Title: PET Imaging Study of α7 and α4β2-nAChR in Schizophrenia: Cognitive Relationships
Brief Title: PET Imaging Study of α7 and α4β2-nAChR in Schizophrenia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study recruitment milestones were not met.
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 202107052
Record Dates: First submitted 2022-06-23; First posted 2022-07-18 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — 3-(1,4-diazabicyclo(3.2.2)nonan-4-yl)-6-fluorodibenzo(b,d)thiophene 5,5-dioxide; 2-(6-fluoro-2,3'-bipyridin-5'-yl)-7-methyl-7-azabicyclo(2.2.1)heptane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Healthy Volunteers (Experimental): Visit 3: (ASEM/AZAN) Blood draw for DNA, PET scan/art line Visit 3: (ASEM only) Blood draw for DNA, PET scan/art line Visit 4: (ASEM only) PET scan/art line
  Interventions: Drug: [18F]ASEM; Drug: [18F]AZAN
- Schizophrenia (ari, brex, risp) (Experimental): Visit 3: (ASEM/AZAN) Blood draw for DNA, PET scan/art line Visit 3: (ASEM only) Blood draw for DNA, PET scan/art line Visit 4: (ASEM only) PET scan/art line
  Interventions: Drug: [18F]ASEM; Drug: [18F]AZAN
- Schizophrenia (olanz) (Experimental): Visit 3: (ASEM/AZAN) Blood draw for DNA, PET scan/art line Visit 3: (ASEM only) Blood draw for DNA, PET scan/art line Visit 4: (ASEM only) PET scan/art line 2-wk Titration, 3-wk steady state
  Interventions: Drug: [18F]ASEM; Drug: [18F]AZAN
- Schizophrenia (no med) (Experimental): Visit 3: (ASEM/AZAN) Blood draw for DNA, PET scan/art line Visit 3: (ASEM only) Blood draw for DNA, PET scan/art line Visit 4: (ASEM only) PET scan/art line 2-wk Titration, 3-wk steady state
  Interventions: Drug: [18F]ASEM; Drug: [18F]AZAN

INTERVENTIONS:
Drug: [18F]ASEM — [18F]ASEM demonstrated excellent imaging properties, as was recently confirmed by others. [18F]ASEM is the 1st validated α7 human PET radiotracer to examine α7-nAChR characteristics in the living brain of SCZ patients. Previous α7 studies in the SCZ literature were done using brains harvested post-mortem, and under variable storage conditions. The proposed studies will also determine α4β2-nAChR [18F]AZAN binding characteristics in the same subjects who complete α7-nAChR PET studies with [18F]ASEM, which will be highly significant for understanding these receptors in SCZ.
Drug: [18F]AZAN — The most widely used PET radioligand for human imaging of α4β2-nAChR is 2-[18F]FA. Because 2-[18F]FA exhibits very slow brain kinetics, the investigators developed [18F]AZAN, a highly α4β2 specific tracer with optimal brain kinetics. Therefore, the proposed studies will utilize [18F]AZAN to determine α4β2-nAChR [18F]AZAN binding characteristics in the same subjects who complete α7-nAChR PET studies with [18F]ASEM, which will be highly significant for understanding these receptors in SCZ.

SUMMARY:
The purpose of this research is to use specialized brain imaging techniques, Positron Emission Tomography (PET) scan and Magnetic Resonance Imaging (MRI), to learn more about the brain chemistry, e.g., how neurotransmitters and receptors in the brain function in people with schizophrenia compared to healthy controls.

DETAILED DESCRIPTION:
Abnormalities in brain chemistry can be responsible for the hallucinations and delusions; thus, by treating these abnormalities, physicians can reduce symptoms of schizophrenia. In this study, investigators aim to examine the characteristics of two investigational radiotracers, [18F]AZAN and [18F]ASEM, in the brains of people with schizophrenia and healthy controls. Radiotracers are drugs in which one or more atoms are "labeled" with a small amount of radioactivity that allows investigators to see how the drug works in humans using PET and MRI brain imaging techniques.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for Healthy Subjects

* Between 18-55 years old (inclusive)men and women.
* Black/African-American or non Hispanic White/Caucasian
* Healthy as determined by medical history, physical examination, clinical laboratory test results, vital signs, and ECG within the reference ranges for the population or results within acceptable deviations that are not clinically significant as determined by study physician.
* Have sufficient arterial or venous access, as determined by Interventional neuroradiologist or anesthesiologist.
* Able to sign written informed consent and to comply with the study restrictions.
* No DSM-5diagnosis on axes I, II, III, and no currently active psychiatric diagnoses or substance use disorders as determined by [SCID]
* If Tobacco or Nicotine user-willing to abstain from products at least 3 hours prior to all PET scans until completion of the scan.

Inclusion Criteria for Patients with Schizophrenia

* Subjects with known chronic SCZ or acute psychotic episodes where suspicion of SCZ is high
* Patients who are drug naïve or nonadherent based on patient report or collateral information OR: a. Subjects on stable (3-months) doses of antipsychotics including risperidone, aripiprazole, ( Part 1 ) Note: if the results of Part 2 ( Aim 4 ) support the null hypothesis for olanzapine effects then investigators will include subjects with schizophrenia on chronic olanzapine. b. Subjects off and then on olanzapine only ( Part 2 )
* 3.18-55 years old (inclusive).
* 4.Male and female subjects meeting DSM-5 diagnostic criteria for a schizophrenia spectrum disorder, verified by SCID-1/P and schizophreniform (<1 year of symptoms5.Black/African-American or non-hispanic White/Caucasian

Exclusion Criteria:

Exclusion Criteria for Healthy Subjects

* Are currently enrolled in or discontinued within the last 30 days from a clinical trial involving an investigational drug or device (other than the study drug) or are currently enrolled in any other type of medical research.
* Have participated in other research protocols specifically regulated under 21 CFR 361.1 in the last year such that radiation exposure would exceed the annual limits.
* Pregnant or nursing women.
* History of head trauma with prolonged loss of consciousness (>10 minutes) or any neurological condition including stroke or seizure (excluding childhood febrile seizure) or history of migraine headache.
* Abnormal vital signs, ECG or clinical laboratory evaluations which are considered clinically significant by the clinical investigator.
* Suffer from claustrophobia and would be unable to undergo MRI or PET scanning.
* Clinically significant abnormal MRI.
* Subject has implanted or embedded metal objects, prostheses, or fragments in the head or body that would present a risk during the MRI scanning procedure, or have worked with ferrous metals either as a vocation or hobby (for example, as a sheet metal worker, welder, or machinist) in such a way that might have led to unknown, indwelling metal fragments that could cause injury if they moved in response to placement in the magnetic field.
* Currently uses prescription medications, over-the-counter drugs or herbal remedies such as St. Johns Wort) which cannot be discontinued 14 days (or <5 half-lives, whichever is longer), prior to the PET scan and throughout the study. Exceptions include daily multiple vitamins.
* Currently a user (including "recreational use") of any illicit drugs or alcohol abuse, or has a positive drug screen.
* Patients undergoing active use of medications that would influence radiotracer binding, including certain 5-HT3 antiemetics, acetylcholine (ACh) receptor agonists (nicotine) or antagonists, and acetylcholinesterase inhibitors.
* History of substance use disorder (DSM-V); or positive alcohol breath test.
* Are currently experiencing neuropsychiatric illness or severe systemic disease based on history and physical exam.

Exclusion Criteria for Patients with Schizophrenia

* Are currently enrolled in or discontinued within the last 30 days from a clinical trial involving an investigational drug or device (other than the study drug) or are currently enrolled in any other type of medical research.
* Have participated in other research protocols specifically regulated under 21 CFR 361.1 in the last year such that radiation exposure would exceed the annual limits.
* Pregnant or nursing women.
* Patients undergoing active use of medications that would influence radiotracer binding, including certain 5-HT3 antiemetics, acetylcholine (ACh) receptor agonists (nicotine) or antagonists, and acetylcholinesterase inhibitors.
* History of head trauma with prolonged loss of consciousness (>10 minutes) or any neurological condition including stroke or seizure (excluding childhood febrile seizure) or history of migraine headache.
* Abnormal vital signs, ECG or clinical laboratory evaluations which are considered clinically significant by the clinical investigator.
* Suffer from claustrophobia and would be unable to undergo MRI or PET scanning.
* Clinically significant abnormal MRI.
* Subject has implanted or embedded metal objects, prostheses, or fragments in the head or body that would present a risk during the MRI scanning procedure, or have worked with ferrous metals either as a vocation or hobby (for example, as a sheet metal worker, welder, or machinist) in such a way that might have led to unknown, indwelling metal fragments that could cause injury if they moved in response to placement in the magnetic field.
* Active substance or alcohol use disorder (including "recreational use") of any illicit drugs meeting criteria for current substance use disorder
* Any subject who has a positive Urine Drug Screen test unless in the Investigator's (Principal Investigator or Sub-Investigator) documented opinion, the positive test does not signal a clinical condition that would impact the safety of the subject or interpretation of the trial results.
* Any subject who has an Alcohol Breathalyzer test result deemed positive by the Investigator (Principal Investigator or Sub-Investigator unless in the Investigator's (Principal Investigator or Sub-Investigator) documented opinion, the positive test does not signal a clinical condition that would impact the safety of the subject or interpretation of the trial results.
* Current treatment with clozapine.
* Current treatment with typical antipsychotics, but not haloperidol.
* Current treatment with antiemetic or smoking cessation medications.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 117 (Actual)
Dates: Start 2022-08-18 (Actual); Primary Completion 2025-01-07 (Actual); Study Completion 2025-01-07 (Actual)

PRIMARY OUTCOMES:
Receptor binding of [18F] ASEM-PET to nicotinic brain receptors (α7-nAChRs) in adults ages 18-55 year with SCZ vs. matched controls. | 60-74 days
  The Primary Outcome Measure is volume of distribution (VT, represented as ml of plasma/cm^3 of tissue) of alpha-7 nicotinic receptors (α7-nAChR) bound to by the [18F]ASEM radio tracer in the brain, comparing VT in people with SCZ with VT in otherwise healthy adults matched for all demographics (smoking status, age, sex, race/genotype, parental education).
Receptor binding of [18F]AZAN to α4β2 nicotinic acetylcholine receptors (α4β2-nAChR) in adults ages 18-55 years with SCZ vs. matched controls. | 60-74 days
  The Primary Outcome Measure is volume of distribution (VT, represented as ml of plasma/cm^3 of tissue) of α4β2 nicotinic acetylcholine receptors (α4β2-nAChR) bound to by the [18F]AZAN radio tracer in the brain, comparing % receptor occupancy in people with SCZ with VT in otherwise healthy adults matched for all demographics (smoking status, age, sex, race/genotype, parental education).
Relationship between α7-nAChR receptor binding VT and negative symptoms in adult patients ages 18-55 yrs with SCZ. | 60-74 days
  The Primary Outcome Measure is the main effect of α7-nAChR receptor volume of distribution (VT, represented as ml of plasma/cm^3 of tissue) on negative symptoms as measured by the negative symptom sub-scale of the Positive and Negative Symptoms Scale (PANSS) in SCZ patients.
Relationship between α4β2-nAChR receptor binding VT and negative symptoms in adult patients ages 18-55 yrs with schizophrenia (SCZ). | 60-74 days
  The Primary Outcome Measure is the main effect of α4β2-nAChR volume of distribution (VT, represented as ml of plasma/cm^3 of tissue) and the negative symptom sub-scale score of the Positive and Negative Symptoms Scale (PANSS) in SCZ.
Relationship between α7-nAChR receptor binding VT and cognitive symptoms, as measured by the Stroop Color-Word Interference Test in SCZ vs. matched controls. | 60-74 days
  The Primary Outcome Measure is the comparison of the main effect of receptor volume of distribution (VT, represented as ml of plasma/cm^3 of tissue) on the Stroop Color-Word Interference Task score in SCZ vs. matched controls.
Relationship between α4β2-nAChR receptor binding VT and cognitive symptoms, as measured by the Stroop Color-Word Interference Task in SCZ vs. matched controls. | 60-74 days
  The Primary Outcome Measure is comparison of the main effect of volume of distribution (VT, represented as ml of plasma/cm^3 of tissue) on the Stroop Color-Word Interference Test score between SCZ patients and matched controls.
Relationship between α7-nAChR receptor binding VT and performance on the Spatial Attention Resource Allocation Task (SARAT) in SCZ vs. matched controls. | 60-74 days
  The Primary Outcome Measure is comparison of the main effect of volume of distribution (VT, represented as ml of plasma/cm^3 of tissue) on the Spatial Attention Resource Allocation Task (SARAT) in SCZ vs. matched controls.
Relationship between α4β2-nAChR receptor binding VT and performance on the Spatial Attention Resource Allocation Task (SARAT) in SCZ vs. matched controls. | 60-74 days
  The Primary Outcome Measure is comparison of the main effect of volume of distribution (VT, represented as ml of plasma/cm^3 of tissue) on the Spatial Attention Resource Allocation Task (SARAT) score in SCZ vs. matched controls.
Relationship between α4β2/α7-nAChR receptor binding VT and cognitive functioning, as measured by the Spatial Attention Resource Allocation Task (SARAT) in SCZ vs. matched controls. | 60-74 days
  The Primary Outcome Measure is the comparison of the interaction between α4β2/α7-nAChR volume of distribution (VT, represented as ml of plasma/cm^3 of tissue) and the Spatial Attention Resource Allocation Task (SARAT) score in SCZ vs. matched controls.
Relationship between α4β2/α7-nAChR receptor binding VT and cognitive functioning, as measured by the Calibrated Neuropsychological Normative Scale (CNNS) score in SCZ vs. matched controls. | 60-74 days
  The Primary Outcome Measure is the comparison of the interaction between α4β2/α7-nAChR volume of distribution (VT, represented as ml of plasma/cm^3 of tissue) and the Calibrated Neuropsychological Normative Scale (CNNS) score in SCZ vs. matched controls.

SECONDARY OUTCOMES:
Relationship between α4β2/α7-nAChR VT and tobacco use disorder in SCZ patients who are smokers vs. non-smoker SCZ patients treated with olanzapine. | 60-74 days
  The Primary Outcome Measure is the relationship between α4β2/α7-nAChR (VT, represented as ml of plasma/cm^3 of tissue) and smoking status in SCZ taking olanzapine who smoke tobacco.
Relationship between the single nucleotide polymorphism (SNP) CHRNA7 rs3087454 and race in SCZ vs. matched controls. | 60-74 days
  The Primary Outcome Measure is the correlation between CHRNA7 rs3087454 and and race (non-Hispanic Caucasians and African Americans) in SCZ vs. matched controls.

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
Plan to share according to NIH guidelines
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code